CLINICAL TRIAL: NCT06999291
Title: Evaluation of Ovarian Reserve in Critically Ill Patients Followed in the Intensive Care Unit
Brief Title: Ovarian Reserve in Intensive Care Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Emine Yilmaz Guler, Principal Investigator, Haseki Training and Research Hospital
Other Study IDs: OR-2024
Record Dates: First submitted 2025-05-07; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Anti-Mullerian Hormone Deficiency
MeSH Terms: interventions — Injury Severity Score

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- internal intensive care: Patients hospitalized in intensive care for internal reasons
  Interventions: Behavioral: Glaskow coma scala, The Acute Physiology and Chronic Health Evaluation System- APACHE, Injury Severity Score- ISS)
- surgical intensive care: Patients hospitalized in intensive care for surgical reasons
  Interventions: Behavioral: Glaskow coma scala, The Acute Physiology and Chronic Health Evaluation System- APACHE, Injury Severity Score- ISS)
- Outpatient clinic patients: Healthy female patients admitted to gynecology outpatient clinic
  Interventions: Behavioral: Glaskow coma scala, The Acute Physiology and Chronic Health Evaluation System- APACHE, Injury Severity Score- ISS)

INTERVENTIONS:
Behavioral: Glaskow coma scala, The Acute Physiology and Chronic Health Evaluation System- APACHE, Injury Severity Score- ISS) — The uterus, endometrium and ovarian characteristics, endometrial thickness, ovarian follicle number and ovarian volume parameters, hormone panel (FSH, LH, E2, AMH), cortisol, prolactin and thyroid function tests routinely examined for ovarian reserve will be evaluated in the study.

SUMMARY:
Gastrointestinal, pulmonary, nephrological, cardiac, neurologic and psychological effects in critically ill patients followed in the intensive care unit have been shown in the literature. However, the effects on ovarian reserve in these patients have not been sufficiently investigated and studies investigating this issue are limited in the literature. The synthesis, release frequency and amplitude of reproductive hormones change under stress. In addition, changes in ovarian homeostasis affect ovarian reserve. The aim of this study was to evaluate ovarian reserve in critically ill patients followed up in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years of age
* Female patients followed in the intensive care unit for more than 24 hours for internal or surgical reasons,
* Women whose ovarian reserve is being evaluated,

Exclusion Criteria:

* Previous ovarian surgery, endometriosis, endometrioma,
* History of chemotherapy, radiotherapy,
* Ovarian cyst, malignancy and other ovarian pathologies,
* Women with single ovary,
* Women receiving hormone therapy,
* Polycystic ovary syndrome,
* Surgical intervention within the last 6 months,
* History of drug, alcohol, substance use,
* Women in pregnancy, puerperium, lactation,
* History of vaccination within the last 6 months

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: a group of healthy women without any disease and a group of patients hospitalized in intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
ovarian follicle count | 24 hour
  Ovarian reserve will be checked with ultrasound

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kayambankadzanja RK, Schell CO, Gerdin Warnberg M, Tamras T, Mollazadegan H, Holmberg M, Alvesson HM, Baker T. Towards definitions of critical illness and critical care using concept analysis. BMJ Open. 2022 Sep 5;12(9):e060972. doi: 10.1136/bmjopen-2022-060972. PMID 36606666
- [Result] Moolhuijsen LME, Visser JA. Anti-Mullerian Hormone and Ovarian Reserve: Update on Assessing Ovarian Function. J Clin Endocrinol Metab. 2020 Nov 1;105(11):3361-73. doi: 10.1210/clinem/dgaa513. PMID 32770239